CLINICAL TRIAL: NCT00000989
Title: A Controlled, Randomized Phase II Study of the Safety and Efficacy of Combined Therapy With Ganciclovir and Granulocyte-Macrophage Colony Stimulating Factor Versus Ganciclovir Alone for the Treatment of Sight-Threatening Cytomegalovirus Retinitis in AIDS Patients
Brief Title: The Safety and Effectiveness of Ganciclovir Used Alone or in Combination With Granulocyte-Macrophage Colony Stimulating Factor in the Treatment of Cytomegalovirus (CMV) of the Eye in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Schering-Plough (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 073; 11047 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Ganciclovir; Drug Evaluation; Drug Therapy, Combination; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; sargramostim; Ganciclovir

INTERVENTIONS:
Drug: Zidovudine
Drug: Sargramostim
Drug: Ganciclovir

SUMMARY:
AMENDED: To evaluate the effect of sargramostim ( GM-CSF ) on modulating the granulocytopenia associated with concomitant DHPG and AZT therapy ( Phase B ), in terms of time to development of granulocytopenia as defined by an absolute neutrophil count ( ANC ) less than or equal to 750 cells/mm3.

Original design: To determine if granulocyte-macrophage colony-stimulating factor ( GM-CSF ) is helpful in preventing the decreased numbers of white blood cells (infection-fighting cells) associated with ganciclovir ( DHPG ) therapy and to determine if GM-CSF can be safely used in AIDS patients with cytomegalovirus ( CMV ) retinitis.

AMENDED: In ACTG 004, among 11 AIDS patients with CMV infection receiving DHPG maintenance therapy (5 mg/kg, 5x/week) with stable white blood cells (WBC)/absolute neutrophil counts (ANC) 7 (64 percent) required dose reduction or discontinuation of both antiviral medications due to granulocytopenia when AZT (600 mg/day) was added. A mean nadir ANC of 717 cells/ml was reached at a mean of 5 weeks of concomitant DHPG/AZT therapy in these patients. While recovery of depressed ANC occurred following discontinuation of study medications, progressive CMV infection (most commonly retinitis) occurred in 19 of 40 patients and seemed to be associated with DHPG therapy interruption. Only 3 of 40 patients were able to tolerate the complete 16 week study duration of DHPG/AZT. Pharmacokinetic studies of co-administration of DHPG and AZT revealed no significant drug-drug interactions. The study investigators concluded that the main, treatment limiting toxicity of combination DHPG/AZT therapy is granulocytopenia and that many patients treated on this study developed intercurrent OIs or staphylococcal septicemia. In order to determine whether patients receiving maintenance DHPG therapy with or without GM-CSF can tolerate concomitant AZT therapy, extended maintenance therapy with the assigned study regimen in combination with AZT will be incorporated into this protocol. Original design: CMV infection causes inflammation of the retina and can lead to permanent blindness. Treatment for CMV retinitis with DHPG has been shown to be effective in halting the progression of retinal disease. During DHPG treatment, however, about 30 to 55 percent of patients develop decreased white blood cell counts. GM-CSF, a naturally occurring human hormone, stimulates the body's bone marrow to produce more white blood cells. Studies with GM-CSF in AIDS patients have shown that it can significantly increase depressed white blood cell counts in these patients.

DETAILED DESCRIPTION:
AMENDED: In ACTG 004, among 11 AIDS patients with CMV infection receiving DHPG maintenance therapy (5 mg/kg, 5x/week) with stable white blood cells (WBC)/absolute neutrophil counts (ANC) 7 (64 percent) required dose reduction or discontinuation of both antiviral medications due to granulocytopenia when AZT (600 mg/day) was added. A mean nadir ANC of 717 cells/ml was reached at a mean of 5 weeks of concomitant DHPG/AZT therapy in these patients. While recovery of depressed ANC occurred following discontinuation of study medications, progressive CMV infection (most commonly retinitis) occurred in 19 of 40 patients and seemed to be associated with DHPG therapy interruption. Only 3 of 40 patients were able to tolerate the complete 16 week study duration of DHPG/AZT. Pharmacokinetic studies of co-administration of DHPG and AZT revealed no significant drug-drug interactions. The study investigators concluded that the main, treatment limiting toxicity of combination DHPG/AZT therapy is granulocytopenia and that many patients treated on this study developed intercurrent OIs or staphylococcal septicemia. In order to determine whether patients receiving maintenance DHPG therapy with or without GM-CSF can tolerate concomitant AZT therapy, extended maintenance therapy with the assigned study regimen in combination with AZT will be incorporated into this protocol. Original design: CMV infection causes inflammation of the retina and can lead to permanent blindness. Treatment for CMV retinitis with DHPG has been shown to be effective in halting the progression of retinal disease. During DHPG treatment, however, about 30 to 55 percent of patients develop decreased white blood cell counts. GM-CSF, a naturally occurring human hormone, stimulates the body's bone marrow to produce more white blood cells. Studies with GM-CSF in AIDS patients have shown that it can significantly increase depressed white blood cell counts in these patients.

AMENDED: Following completion of Phase A, study participants may elect to extend their assigned maintenance therapy (DHPG alone or DHPG/GM-CSF) in combination with AZT therapy (Phase B). GM-CSF dosing will be titrated as above to maintain a target ANC of 2500-5000 cells/mm3. Those patients receiving DHPG/AZT who develop neutropenia (ANC less than 750/ml) on two occasions will begin GM-CSF to maintain a target ANC of 2500-5000 cells/mm3. A similar schedule of clinical, ophthalmologic and laboratory evaluations will be followed in order to determine the efficacy and safety of extended maintenance therapy combined with AZT. Close monitoring of antiviral (CMV, HIV) and immunomodulatory activity will be assessed. This second phase of the study will last for an additional 52 weeks. AMENDED: Extended to 68 weeks. Original design: Patients are hospitalized for a minimum of 7 days to begin treatment for CMV retinitis. They are randomly assigned to one of two groups to receive DHPG either with or without GM-CSF. DHPG is given by intravenous infusion every 12 hours for the first 14 days. DHPG maintenance therapy is then given once a day, 7 days/week for the remaining 14 weeks of the study. For patients in the DHPG with GM-CSF group, the GM-CSF is given by subcutaneous injection for the 16 weeks of the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Maintenance therapy for stable opportunistic infection which is not myelosuppressive.
* Aerosolized pentamidine for prophylaxis of Pneumocystis carinii pneumonia.
* Acyclovir or other appropriate medications for appearance of Herpes simplex virus or Varicella zoster virus infections (after enrollment in study) that require systemic therapy.
* Medications absolutely necessary for the patient's welfare, at discretion of investigator.

Patients must:

* Have a diagnosis of sight-threatening cytomegalovirus (CMV) retinitis and AIDS.
* Have at least one pending culture for cytomegalovirus (CMV) from buffy coat and/or urine prior to study entry or previously documented CMV viremia or viruria within 6 weeks prior to study entry.
* Be capable of giving informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Corneal, lenticular, or vitreal opacification that precludes examination of the fundi, or evidence of other retinopathy other than cotton wool spots.

Concurrent Medication:

Excluded:

* Systemic antiviral therapy except Zidovudine (AZT) which will be added during the extended maintenance phase of the study.
* Foscarnet.
* Treatment for an active AIDS-defining opportunistic infection.
* Any potentially cytotoxic chemotherapeutic agent.

Patients with the following are excluded:

* Corneal, lenticular, or vitreal opacification that precludes examination of the fundi, or evidence of other retinopathy other than cotton wool spots.

Prior Medication:

Excluded within 14 days of study entry:

* Other immunomodulators, biologic response modifiers, or investigational agents.
* Protocol drugs.
* Foscarnet.
* Any potentially cytotoxic chemotherapeutic agent.

Prior Treatment:

Excluded within 14 days of study entry:

* Administration of cytomegalovirus hyperimmune globulin in therapeutic doses.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Study Completion 1992-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hardy WD, Study Chair
Locations (4):
- United States (4):
  - UCLA CARE Center CRS, Los Angeles, California
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina

REFERENCES:
- [Background] Hardy D, et al. Ganciclovir (GCV) and granulocyte-macrophage colony stimulating factor (GM-CSF) vs GCV alone as treatment for cytomegalovirus (CMV) retinitis (ACTG 073). Int Conf AIDS. 1992 Jul 19-24;8(1):Mo5 (abstract no MoA 0005)
- [Background] Hardy D, Spector S, Polsky B, Crumpacker C, van der Horst C, Holland G, Freeman W, Heinemann MH, Sharuk G, Klystra J, et al. Combination of ganciclovir and granulocyte-macrophage colony-stimulating factor in the treatment of cytomegalovirus retinitis in AIDS patients. The ACTG 073 Team. Eur J Clin Microbiol Infect Dis. 1994;13 Suppl 2:S34-40. doi: 10.1007/BF01973600. PMID 7875151
- [Background] Hardy WD. Combined ganciclovir and recombinant human granulocyte-macrophage colony-stimulating factor in the treatment of cytomegalovirus retinitis in AIDS patients. J Acquir Immune Defic Syndr (1988). 1991;4 Suppl 1:S22-8. PMID 1848618